CLINICAL TRIAL: NCT06411301
Title: A Phase I Study to Assess the Tolerability of 225Ac-DOTATATE in Patients With Refractory and Relapsing Multiple Myeloma Expressing Somatostatin Receptors
Acronym: AcTRESS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Jules Bordet Institute (Other)
Collaborators: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-MN-AcTRESS
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma, Refractory; Multiple Myeloma in Relapse; Multiple Myeloma Progression
Keywords: Multiple Myeloma; Somatostatin receptor; Radionuclide therapy; Actinium-225; Targeted alpha therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 225Ac-DOTATATE (Experimental): Dose escalation study to assess the safety and determine the recommended phase II dose, based on time-to-event Bayesian optimal interval design, with a target toxicity rate of 30%. Three dose levels are planned to be evaluated: 5 MBq (starting dose), 7.5 MBq and 10 MBq (maximum dose allowed). The cohort size will be 3, with a maximum of 10 participants within a same dose level, and a maximum of 18 evaluable participants in total. Participants are planned to receive two cycles of intravenous infusion of 225Ac-DOTATATE every 6 weeks (Q6W). Each dose escalation and potential de-escalation step will be decided based on the dose-limiting toxicities (DLT) rate observed during the study treatment period (84 days following the first infusion), in the current dose cohort.
  Interventions: Drug: 225Ac-DOTATATE

INTERVENTIONS:
Drug: 225Ac-DOTATATE — Two intravenous infusions every 6 weeks (Q6W)
  Other Names: RYZ101

SUMMARY:
This study aims to determine the safety and the recommended phase II dose of RYZ101 (actinium-225 labelled DOTA-octreotate (225Ac-DOTATATE)) in participants with refractory and relapsing multiple myeloma (MM) that have received at least 3 prior lines of myeloma therapy. Participants will be selected based on somatostatin receptor (SSTR) positivity assessed by gallium-68 labelled DOTA-octreotate (68Ga-DOTATATE) PET/CT. The response to 225Ac-DOTATATE therapy will also be assessed in the target study population.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent in accordance with institutional guidelines and obtained prior to any study procedure
2. Age of at least 18 years at the time of signing the informed consent
3. Confirmed diagnosis of multiple myeloma according to the Salmon and Durie criteria
4. Have received at least 3 prior lines of myeloma therapy including an immunomodulatory drug, a proteasome inhibitor and an anti-CD38 antibody
5. Must have progressed on their last line of myeloma therapy
6. Biologically active (relapsing or refractory) and measurable disease as defined by at least one of the following:

   * Serum M-protein ≥ 0.5 g/dL by serum protein electrophoresis (SPEP) or, for immunoglobulin (Ig) A myeloma, by quantitative IgA
   * Urinary M-protein of at least 200 mg/24 hours by urine protein electrophoresis
   * Serum free light chain (FLC) ≥ 100 mg/L, provided that FLC ratio is abnormal
   * If SPEP is felt to be unreliable for routine M-protein measurement (example, for IgA or IgD MM), then quantitative Ig levels by nephelometry or turbidimetry are acceptable
7. Estimated life expectancy above 6 months
8. Eastern Cooperative Oncology Group performance status ≤ 1
9. Bone marrow aspiration and biopsy sample available within 30 days prior study enrolment (optional under the subject agreement)
10. Baseline PET/CT imaging scans defined by:

    * 68Ga-DOTATATE PET/CT-positive imaging with target lesions, defined as unequivocal tumoral uptake higher than the maximum standardized uptake value of the femoral bone marrow background
    * All 18F-FDG PET/CT-avid lesions must be SSTR-positive, as defined above
11. Adequate renal function as measured by renal scintigraphy scans and evidenced by creatinine clearance (CrCl) ≥60 mL/min/1.73m^2
12. Adequate hematologic function defined by the following laboratory results:

    * Hemoglobin concentration ≥5.0 mmol/L (≥8.0 g/dL)
    * Total white blood cell count ≥1.5 × 103/mm^3
    * Absolute neutrophil count ≥1000 cells/µL (≥1000 cells/mm^3)
    * Platelets count >100 × 10^9/L (100 × 10^3/mm^3)
13. Adequate hepatic function defined by the following laboratory results:

    * Aspartate aminotransferase and alanine aminotransferase ≤2.5 × upper limit of normal (ULN) (or ≤5 × ULN if presence of liver metastases)
    * Total bilirubin ≤3 × ULN
    * Serum albumin ≥3.0 g/dL
14. Adequate coagulation function, defined by international normalized ratio or prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN, unless subject is receiving anticoagulant therapy and PT or aPTT is within therapeutic range of intended use of anticoagulants
15. For women of childbearing potential (WOCBP):

    * Negative serum pregnancy test within 48 hours prior to the first dose of study treatment
    * Agreement to use barrier contraception and a second form of highly effective contraception (Clinical Trials Facilitation Group (CTFG) 2020) while receiving study treatment and for 7 months following their last dose of study treatment
16. Sexually active male subjects must use a condom during intercourse while receiving study treatment and for at least 120 days after the last dose of the study drug and should not father a child during this period

    * Male study subjects whose sexual partners are WOCBP must also agree to use a second form of highly effective contraception (CTFG 2020) while receiving study treatment and for at least 4 months following their last dose
    * Vasectomized men are also required to use a condom during intercourse, including with a male partner

Exclusion Criteria:

1. Massive bone marrow infiltration on the baseline 68Ga-DOTATATE PET/CT scan
2. History of hypersensitivity or allergy to 225Ac, 68Ga, octreotate, or any of the excipients of DOTATATE imaging agents
3. Use of anticancer agents within the following intervals prior to the first dose of study drug:

   * Chemotherapy: within <6 weeks
   * Small molecule inhibitors: within <4 weeks
   * Biological agents: within <7 days or <5 half-lives
4. Prior external beam radiotherapy on more than 25% of bone marrow
5. Prior participation in any interventional clinical study within 30 days prior to first dose of study drug
6. Have a history of primary malignancy within the past 3 years other than (1) MM; (2) adequately treated carcinoma in situ or non-melanoma carcinoma of the skin; (3) any other curatively treated malignancy that is not expected to require treatment for recurrence during participation in the study, or (4) an untreated cancer on active surveillance that may not affect the subject's survival status for ≥3 years based on clinician assessment/statement
7. Any toxicities from prior treatments that have not recovered to CTCAE Grade ≤1 at baseline, except for alopecia
8. Significant cardiovascular disease, defined as:

   * New York Heart Association (NYHA) Class ≥II heart failure
   * Known left ventricular ejection fraction <50%
   * History of myocardial infarction, acute coronary syndrome, or coronary angioplasty/stenting/bypass within the last 6 months
   * QT interval corrected for heart rate using Fridericia's formula >470 ms, demonstrated by the average value of 3 consecutive electrocardiograms
9. Resistant hypertension, defined as persistent uncontrolled blood pressure >140/90 mmHg (diastolic/systolic) while on optimal doses of at least 3 antihypertensive medications with 1 being a diuretic
10. Uncontrolled diabetes mellitus as defined by hemoglobin A1C >8%
11. Impossibility to discontinue corticoids administration at a therapeutic level (total dose of 160 mg of dexamethasone or equivalent) two weeks prior dosing of study drug
12. Pregnancy or lactation
13. Any known or underlying medical, psychiatric disease/condition, and/or social situations that, in the opinion of the investigator, would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of 225Ac-DOTATATE | First 84 days following first 225Ac-DOTATATE injection
  Incidence and severity of adverse events (AEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Recommended phase II dose of 225Ac-DOTATATE | First 84 days following first 225Ac-DOTATATE injection
  Rate incidence of dose-limiting toxicities (DLT)

SECONDARY OUTCOMES:
Clinical activity of treatment with 225Ac-DOTATATE | First 84 days following first 225Ac-DOTATATE injection
  Overall response according to the International Myeloma Working Group (IMWG) response criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Jules Bordet Institute, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No